CLINICAL TRIAL: NCT05798962
Title: Cellular Mechanisms Involved in Pathology Following Musculo-tendinous Injuries
Brief Title: Cellular Mechanisms Involved in Muscle Pathology
Status: Recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Monika Lucia Bayer, Senior Researcher, Bispebjerg Hospital
Other Study IDs: P162
Record Dates: First submitted 2023-02-27; First posted 2023-04-05 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Muscle Strain, Lower Leg; Muscle Strained Thigh; Achilles Tendon; Laceration; Fatty Degeneration
MeSH Terms: conditions — Sprains and Strains; Lacerations; Fatty Liver | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 biopsy from the pathological skeletal muscle
  1 biopsy from the contralateral, healthy muscle (i.e. the healthy muscle corresponding to the injured muscle)
  1 biopsy from the healthy, uninjured vastus lateralis muscle
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute muscle strain: Subjects with an acute muscle strain (within 14 days post injury) in either the hamstrings or the calf muscles
  Interventions: Procedure: Biopsies
- Chronic muscle strain: Subjects with a chronic muscle strain more than 6 months prior to inclusion in either the hamstrings or the calf muscles
  Interventions: Procedure: Biopsies
- Achilles tendon rupture: Subjects with a full Achilles tendon rupture more than 12 months prior to inclusion
  Interventions: Procedure: Biopsies

INTERVENTIONS:
Procedure: Biopsies — Biopsies from the pathological muscle and healthy, unaffected muscle

SUMMARY:
The overall purpose of this proposed study is the understanding of cellular mechanisms involved in the pathologic fatty degeneration of muscle. Fatty infiltration in skeletal muscle is observed following sports injuries such as muscle strain injuries and Achilles tendon rupture. It is also observed in the degenerative state after rotator cuff tears as well as in the aging process. While fatty degeneration of skeletal muscle occurs in many different conditions and is known to decrease muscle function, the cellular processes involved in fatty infiltration have not been investigated in human muscle.

Hypotheses:

1. There is a high amount of fibro-adipogenic progenitors (FAPs) with an adipogenic pattern in pathologic skeletal muscle following a muscle strain injury and a full Achilles tendon rupture. We hypothesize that there is an increased number of FAPs with an adipogenic signature already in the acute phase after a strain injury, but a significantly higher number in the chronic stage as well as in the muscle following an Achilles tendon rupture.
2. Mechanical cues are a major driver of the phenotypic drift of FAPs. The lack of mechanical stimuli initiates the adoption of an adipogenic pathway in naïve FAPs, whereas naïve FAPs exposed to mechanical stimuli will maintain their undifferentiated phenotype.
3. The adherence of FAPs to a soft material will activate the adoption of an adipogenic phenotype, whereas a stiff material will favor a more fibrotic phenotype in naïve FAP's isolated from healthy skeletal muscle.

DETAILED DESCRIPTION:
Skeletal muscle strain injury is one of the most common sports injuries, which is caused by excessive tensile strain of the muscle and affects the region where muscle fascicles insert into the connective tissue (aponeurosis). It is therefore not an injury solely affecting skeletal muscle, but the skeletal muscle-aponeurosis interface. Having sustained one strain injury increases the risk of re-injury substantially, changes the biomechanics of the involved muscle and leads to a significantly enlarged aponeurosis. Recently, the investigators have discovered the accumulation of ectopic fat in the intra-fascicular space and within myofibrils. The built-up of ectopic fat in skeletal muscle is a degenerative state and has mostly been described for rotator cuff injuries where it is associated with worse shoulder functional scores. At the same time, the investigators have observed a high cellularity in the pathologic muscle-aponeurosis following strain injuries, but it is not known what cell types these cells are. It seems therefore likely that at least some of the cells are Fibro/adipogenic progenitors (FAPs), which contribute to the fat accumulation in strain injured muscles and that fat accumulation might be a factor contributing to the high risk of recurrent injuries, as well as other medical problems such as pain and decreased function often described long time after a strain injury.

Another common injury of the lower leg is the full Achilles tendon rupture. Recent data show that patients have long-term impairments in the injured leg when compared to the non-injured side. Also after full Achilles tendon ruptures, fatty degeneration of the muscles in the calf has been reported and has been linked to poor patient outcome. Recently, the investigators have observed fatty infiltration of calf muscles in patients following Achilles tendon rupture, which might lead to a decrease in muscle function and thereby to a poor patient outcome.

Despite the high prevalence of muscle strain injuries, very little is known about the cellular mechanisms following a strain injury. In addition, the literature on the cellular composition and alterations following Achilles tendon ruptures is scarce. A decade ago, a group of cells named fibro/adipogenic progenitors (FAPs) have been identified in the interstitial space of skeletal muscle based on the presence of stem cell antigen 1+, CD34+, Platelet Derived Growth Factor Receptor α (PDGFR α)+ . Aside from their supporting activity in muscle regeneration, FAPs have the potential to adopt an adipogenic or profibrotic phenotype. Despite the high incidence, it has not been studied whether the traumatic injury and the subsequent biomechanical changes in the skeletal muscle and associated connective tissue following strain injuries or Achilles tendon rupture activate FAPs, and how these cells contribute to the fatty accumulation in the skeletal muscle.

Hypotheses:

1. There is a high amount of fibro-adipogenic progenitors (FAPs) with an adipogenic pattern in pathologic skeletal muscle following a muscle strain injury and a full Achilles tendon rupture. The investigators hypothesize that there is an increased number of FAPs with an adipogenic signature already in the acute phase after a strain injury, but a significantly higher number in the chronic stage as well as in the muscle following an Achilles tendon rupture.
2. Mechanical cues are a major driver of the phenotypic drift of FAPs. The lack of mechanical stimuli initiates the adoption of an adipogenic pathway in naïve FAPs, whereas naïve FAPs exposed to mechanical stimuli will maintain their undifferentiated phenotype.
3. The adherence of FAPs to a soft material will activate the adoption of an adipogenic phenotype, whereas a stiff material will favor a more fibrotic phenotype in naïve FAP's isolated from healthy skeletal muscle.

To test this, the investigators will take small tissue samples from the injured area in either the acute phase (subject group A) or the chronic phase (subject group B) after a strain injury as well as from the muscle tissue of individuals who had a full Achilles tendon rupture at least a year prior to inclusion (subject group C). In all three groups, the investigators will also take a small tissue sample from the same muscle as the injured one on the healthy side. In addition, a larger muscle biopsy from the contralateral healthy vastus lateralis muscle is taken to compare the cellular composition and the cellular profile between the pathologic skeletal muscle-aponeurosis and a healthy skeletal muscle.

To test the importance of mechanical stimuli, isolated muscle cells will be sorted with Fluorescence Activated Cell Sorting (FACS) and cultured in vitro thereafter. The investigators particularly focus on culture under static and dynamic tension and in the de-tensioned state.

An alpha level of 0.05 will be considered significant. Based on previous data, 10 participants will be recruited for each group, enabling the investigators to detect an estimated doubling of FAPs in the injured muscles (primary outcome). Power analysis for the primary outcome resulted in n=4 for each group (α=0.05, β=0.80, CV=72.4%), which the investigators consider to be clinically relevant. The investigators plan to include 10 participants in each group to have sufficient biopsy material from 5 individuals for single nuclei RNA sequencing and 5 biopsies for fluorescence-activated cell sorting and the subsequent in vitro studies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, male and female, with an acute muscle strain injury (<14 days post injury) in the calf or hamstring muscles (group 1). Pathological changes visible on an ultrasound scan as hypoechoic areas.
* 18 years and older, male and female, with a chronic muscle strain injury (> 6 months prior to inclusion) in the calf or hamstring muscles (group 2), sequela including recurrent strain injuries, pain and/ or decrease in muscle function. Pathological changes visible on an ultrasound scan as hypo-/ hyperechoic areas.
* 18 years and older, male and female, with a full Achilles tendon rupture (> 1 year prior to inclusion) with pathological changes: Fatty degeneration visible on an ultrasound scan (group 3).

Exclusion Criteria:

* Type I and II Diabetes, Connective tissue and/or rheumatic diseases, or any observed organ dysfunctions
* Daily smoking
* Persons with daily intake of non-steroidal anti-inflammatory drugs (NSAIDs) within three months prior to time of contact
* Allergic reactions to local anesthesia
* Use of anticoagulant treatment
* Needle phobia
* Any drug or alcohol abuse now or in the past
* The absence of any pathological changes visible on an ultrasound scan as hypo-/ hyperechoic areas (group 1 and 2)
* The absence of any pathological changes (fatty degeneration) in either the gastrocnemius or the soleus muscle visible on an ultrasound scan (Subject group 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals with an acute or previous muscle strain injury or a previous Achilles tendon rupture
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Presence and number of Fibro-adipogenic progenitors | 2 years: Sampling and analyses
  Determination of the number and the phenotypic appearance of fibro-adipogenic progenitors in the injured compared to the healthy muscle

SECONDARY OUTCOMES:
Cell cluster analysis | 2 years: Sampling and analyses
  Analysis of cell clusters present in the injured compared to the healthy muscle by single nuclei RNA sequencing
Importance of mechanical stimuli for Fibro-adipogenic progenitors | 2 years: Sampling and analyses
  Importance of mechanical stimuli on the phenotypic drift of fibro-adipogenic progenitors ("FAPS". Isolated FAP´s will be subjected to either mechanical stimulation (by using the FlexCell system) or unloading ("FAPs embedded in a free-floating matrix). FAPs will also be cultured on stiff versus soft surfaces to study thereafter the effect of the substrate properties on the phenotypic appearance of FAPs. The phenotypic appearance of FAPs will be tested by qRT-PCR, protein analysis and compared to the well-described effect on phenotypic apprearance of FAPs when subjected to pro-fibrotic or pro-adipogenic differentiation medium.

CONTACTS AND LOCATIONS:
Overall Officials: Monika L Bayer, PhD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Nielsine Nielsen Vej 11, Building 8, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayer ML, Hoegberget-Kalisz M, Jensen MH, Olesen JL, Svensson RB, Couppe C, Boesen M, Nybing JD, Kurt EY, Magnusson SP, Kjaer M. Role of tissue perfusion, muscle strength recovery, and pain in rehabilitation after acute muscle strain injury: A randomized controlled trial comparing early and delayed rehabilitation. Scand J Med Sci Sports. 2018 Dec;28(12):2579-2591. doi: 10.1111/sms.13269. Epub 2018 Aug 16. PMID 30043997
- [Background] Ekstrand J, Walden M, Hagglund M. Hamstring injuries have increased by 4% annually in men's professional football, since 2001: a 13-year longitudinal analysis of the UEFA Elite Club injury study. Br J Sports Med. 2016 Jun;50(12):731-7. doi: 10.1136/bjsports-2015-095359. Epub 2016 Jan 8. PMID 26746908
- [Background] Bayer ML, Hoegberget-Kalisz M, Svensson RB, Hjortshoej MH, Olesen JL, Nybing JD, Boesen M, Magnusson SP, Kjaer M. Chronic Sequelae After Muscle Strain Injuries: Influence of Heavy Resistance Training on Functional and Structural Characteristics in a Randomized Controlled Trial. Am J Sports Med. 2021 Aug;49(10):2783-2794. doi: 10.1177/03635465211026623. Epub 2021 Jul 15. PMID 34264782
- [Background] Gladstone JN, Bishop JY, Lo IK, Flatow EL. Fatty infiltration and atrophy of the rotator cuff do not improve after rotator cuff repair and correlate with poor functional outcome. Am J Sports Med. 2007 May;35(5):719-28. doi: 10.1177/0363546506297539. Epub 2007 Mar 2. PMID 17337727
- [Background] Uezumi A, Fukada S, Yamamoto N, Takeda S, Tsuchida K. Mesenchymal progenitors distinct from satellite cells contribute to ectopic fat cell formation in skeletal muscle. Nat Cell Biol. 2010 Feb;12(2):143-52. doi: 10.1038/ncb2014. Epub 2010 Jan 17. PMID 20081842
- [Background] Uezumi A, Ito T, Morikawa D, Shimizu N, Yoneda T, Segawa M, Yamaguchi M, Ogawa R, Matev MM, Miyagoe-Suzuki Y, Takeda S, Tsujikawa K, Tsuchida K, Yamamoto H, Fukada S. Fibrosis and adipogenesis originate from a common mesenchymal progenitor in skeletal muscle. J Cell Sci. 2011 Nov 1;124(Pt 21):3654-64. doi: 10.1242/jcs.086629. Epub 2011 Nov 1. PMID 22045730